CLINICAL TRIAL: NCT00145652
Title: Phase 3 Study of Recombinant Erythropoetin and Adjuvant I.V. Iron Therapy of Anemic Patients With Lymphoproliferative Disorders
Brief Title: Adjuvant I.V. Iron Therapy During Erythropoetin Treatment of Anemic Patients With Lymphoproliferative Disorders.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sundsvall Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Hedenus; Medical Products Agency; Dnr:151:2003/29970
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2006-09

CONDITIONS: Anemia; Multiple Myeloma; Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: erythropoetin; adjuvant iron therapy; anemia; cancer
MeSH Terms: conditions — Anemia; Multiple Myeloma; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — Ferric Oxide, Saccharated

INTERVENTIONS:
Drug: Neo-Recormon and Venofer

SUMMARY:
This is a multi-center open label, randomized phase-3 study with stratification according to diagnosis and baseline serum-EPO level. The correction of mild or moderate anemia and the effect on iron kinetics by the rHuEPO treatment with or without intravenous iron supplementation in anemic patients with LPD not receiving antineoplastic therapy will be studied. The study will be performed according to the ICH-GCP guidelines. In order to be eligible, the patient must consent in writing that he/she agrees to participate in the study. The patient recruitment period is estimated to be no longer than 18 months.

DETAILED DESCRIPTION:
In this multi-center, randomized, open label phase-3 study, the correction of mild or moderate anemia and the effect on iron kinetics by rHuEPO treatment, with or without intravenous iron treatment, in patients with LPD not receiving antineoplastic therapy will be studied.

LENGTH OF STUDY 16 weeks

NUMBER OF CENTERS 15

NUMBER OF SUBJECTS 66

STRATIFICATION 1. According to diagnosis; CLL and indolent NHL vs. MM. 2. According to level of S-epo > 100 IU/L vs £ 100 IU/L at baseline.

TREATMENT The patients will be randomized to receive 30 000 IU Neorecormon â (epoetin beta) s.c. once / week for 16 consecutive weeks +/- 100mg/week of Venofer â (iron sucrose) from week 0 to 6, followed by one 100mg dose every 2 week from weeks 8 until 14.

If the increase in Hb concentration is less than 10g/L from baseline (week 0) until week 4 weeks, the dose of epoetin beta will be increased to 60 000 IU weekly from week 5.

If the Hb concentration exceeds 140 g/L, the epoetin beta therapy will be suspended. The treatment will be resumed once the Hb concentration falls below 130 g/L. This resumed dose will be 75% of the previous dose (e.g. if the previous dose was 30 000 IU before suspension, the continued dose should be 22 500 IU. If the dose was 60 000 IU before suspension, the dose should be 45 000 IU).

If the level of S-ferritin reaches >1000 ug/L iron sucrose should be suspended until the S-ferritin level falls below 500 ug/L.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma, indolent NHL or CLL
* Anemia of cancer with a Hb concentration within the range ³ 90 - £ 110 g/L measured at two different occasions with at least two weeks interval but inclusion within 4 weeks after the first Hb measurement.
* Age >18 years.
* Informed consent in writing.
* Demonstration of stainable iron in bone-marrow aspirate.

Exclusion Criteria:

* Planned or expected antineoplastic therapy (except systemic low dose maintenance corticosteroids) within the 6 weeks following inclusion.
* Cytostatic or any other antitumor therapy (except systemic low dose maintenance corticosteroids) within 8 weeks before inclusion.
* RBC transfusion within 8 weeks before inclusion.
* RHuEPO treatment within 12 weeks before inclusion.
* Any iron therapy within 4 weeks before inclusion.
* Ongoing infectious disease.
* Active inflammatory disease other than the malignant disease.
* Performance status ³ 3 according to the ECOG scale.
* Folate deficiency (S-folate < 4,5 nmol/L).
* B12 deficiency (S-cobalamin < 145 pmol/L).
* Ongoing haemolysis defined as S-haptoglobin < 0,2 g/L
* Impaired kidney function (S-Creatinine > 175 mmol/L)
* Acute or chronic clinical relevant hepatic dysfunction (S-bilirubin >40 umol/L)
* S-Ferritin >800 ug/L
* Ongoing significant neurological or psychiatric disorders including psychotic disorders or dementia.
* Unstable or uncontrolled disease related to or affecting cardiac function e.g., unstable angina, congestive heart failure (NYHA>Class ll), uncontrolled hypertension (diastolic BP >100 mmHg) and/or uncontrolled cardiac arrhythmia.
* Known history of allergy to any of the study medications or their excipients.
* Concurrent treatment with experimental drugs not approved by Läkemedelsverket.
* Male and female patients with reproductive potential must use an approved contraceptive method (e.g. intrauterine device (IUD), birth control pills or barrier device) during the study and for 3 months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrolment.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66
Dates: Start 2003-12; Study Completion 2005-12

PRIMARY OUTCOMES:
To compare the mean change in hemoglobin (Hb) concentrations from baseline to EOT (End of treatment ) between the two treatment groups.

SECONDARY OUTCOMES:
The percentage of subjects with Hb response defined by an increase in the Hb concentration by at least 20 g/L in the absence of any RBC transfusion.
The time needed to obtain a Hb response.
The fraction of subjects receiving RBC transfusions during the study period.
The dose of rHuEPO used.
The effect on iron-status.
The weekly Hb concentration profile over time.
The frequency and grade of adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hedenus, MD, Principal Investigator — Unaffilitated
Locations (1):
- Michael Hedenus, Sundsvall, Sweden

REFERENCES:
- [Background] Auerbach M, Ballard H, Trout JR, McIlwain M, Ackerman A, Bahrain H, Balan S, Barker L, Rana J. Intravenous iron optimizes the response to recombinant human erythropoietin in cancer patients with chemotherapy-related anemia: a multicenter, open-label, randomized trial. J Clin Oncol. 2004 Apr 1;22(7):1301-7. doi: 10.1200/JCO.2004.08.119. PMID 15051778